CLINICAL TRIAL: NCT05803590
Title: Comparative Effect of Green Tea Versus Chlorhexidine Mouthwash on Plaque Induced Gingivitis In a Group of Egyptian Children: Randomized Clinical Trial
Brief Title: Compare the Effect of Green Tea Mouthwash vs Chlorohexidine Mouthwash in Children With Plaque-induced Gingivitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Abd Elnaser Yehia Fatoh, The Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GT Mouthwash In Children
Record Dates: First submitted 2023-03-08; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Plaque Induced Gingivitis
Keywords: green tea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding of the operator and the patients will not be applicable due to the difference between the used mouthwashes. However, the statistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green Tea Mouthwash ( intervention ) (Active Comparator): Green tea (GT), obtained from the extracts of a small plant, Camelia sinesis, is common worldwide. It is rich in flavonoids such as catechins and various other polyphenols, contributing to its antioxidant and anti-inflammatory properties. Green tea consumption is also associated with lower incidences of diabetes, cardiovascular disease, and obesity. Moreover, its antibacterial property aids in the reduction of bacterial colonization and thereby prevents oral diseases such as gingivitis, periodontal diseases, dental caries, and malodor .
  When used as a mouthwash, green tea preparations can obliterate bad breath by suppressing anaerobic bacteria and eradicating the production of volatile sulfur compounds. There is a lack of critically appraised summaries on the efficacy of green tea mouthwash for promoting dental hygiene .
  Interventions: Drug: Green tea mouthwash; Drug: Chlorhexidine mouthwash
- Chlorhexidine Mouthwash ( control ) (Experimental): Chlorhexidine was developed in 1950 and is the most used anti-plaque agent. However, the long-term usage of chlorhexidine (CHX) is limited by altered taste perception and tooth staining with prolonged usage. Though CHX has been the gold standard mouthwash in controlling plaque formation, its undesirable side effects, such as the enhanced ability of calculus formation, bitter taste, and interference with taste, have inspired a search for alternatives
  Interventions: Drug: Green tea mouthwash; Drug: Chlorhexidine mouthwash

INTERVENTIONS:
Drug: Green tea mouthwash — effictive against caries and periodontal diseases
Drug: Chlorhexidine mouthwash — the gold standard against which other anti-plaque and gingivitis agents are measured

SUMMARY:
This study aims to assess and compare the effect of green tea mouthwash compared to chlorohexidine mouthwash in reducing gingivitis and plaque scores (in terms of plaque index and gingival index) in children with plaque-induced gingivitis.

DETAILED DESCRIPTION:
This study aims to assess and compare the effect of green tea mouthwash compared to chlorohexidine mouthwash in reducing gingivitis and plaque scores (in terms of plaque index and gingival index) in children with plaque-induced gingivitis.

This study will be conducted in the outpatient clinics of the Pediatric Dentistry and Dental Public Health Department - Faculty of Dentistry, Cairo University - Egypt.

Patients attending the outpatient clinic in Pediatric Dentistry and Dental Public health Department - Faculty of Dentistry - Cairo University - Egypt will be screened until the target population is achieved.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 10-14 years.
* Children with a gingival index score of ≥ 1 and a plaque index score of ≥ 1.
* Children in good medical health and free from major oral hard or soft tissue lesions. [Medically fit children (ASA I, II)].
* Children classified as cooperative or potentially cooperative according to Wright's classification of child behavior.
* Children mentally capable of communication.

Exclusion Criteria:

* Parental refusal for participation.
* Children under antibiotics treatment during the last six weeks prior to the study.
* Children wearing fixed or removable orthodontic devices.
* Patients who underwent oral prophylaxis in the last six months.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Gingivitis will be recorded by the Gingival index | one hour
  Gingival Index (GI): (Loe and Sillness Index) records qualitative changes in the gingiva. It scores the marginal and interproximal tissues separately based on 0 to 3. The criteria are:
  0= Normal gingiva.
  1= Mild inflammation - a slight change in color and slight edema but no bleeding on probing. 2= Moderate inflammation - redness, edema, and glazing, bleeding on probing.
  3= Severe inflammation - marked redness and edema, ulceration with the tendency to spontaneous bleeding.
  The bleeding is assessed by gently probing along the wall of the soft tissue of the gingival sulcus. The scores of the four areas of the tooth can be summed and divided by four to give the GI for the tooth. The GI of the individual can be obtained by adding the values of each tooth and dividing by the number of teeth examined. The Gingival Index may be scored for all surfaces or selected teeth or for selected areas of all teeth.

SECONDARY OUTCOMES:
Presence of dental plaque will be recorded by the Plaque index | one hour
  Plaque Index (PI): (Sillness and Loe Index) is an index for estimating the status of oral hygiene by measuring dental plaque that occurs in the areas adjacent to the gingival margin (the gingival one-third of the teeth). It can be used on all teeth or selected teeth. It is used on all four surfaces (M, B, D, L). The criteria are:
  0= No plaque.
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth, which can not be seen with the naked eye. But only by using disclosing solution or using a probe.
  2. Moderate accumulation of deposits within the gingival pocket, on the gingival margin and/ or adjacent tooth surface, which can be seen with the naked eye.
  3. Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.

OTHER OUTCOMES:
Patient Satisfaction using a questionnaire | one hour
  The participants will be asked to fill in at the end of the observation period a questionnaire to indicate on a 0 to 3 scale (0, disagree; 1 slightly disagree; 2, slightly agree; 3, agree) his/her level of agreement to nine statements concerning the mouthwashes under investigation regarding safety, tolerability, pleasantness, and performance.